CLINICAL TRIAL: NCT06385717
Title: Multicenter Cohort Study of Chemo-radiotherapy After Endoscopic Submucosal Dissection for High-risk Early-stage Esophageal Cancer
Brief Title: Multicenter Cohort Study of ESD and Chemo-radiotherapy for High-risk Early-stage Esophageal Cancer
Acronym: ESCORT
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ZhejiangU
Record Dates: First submitted 2024-04-11; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Esophagus Cancer
Keywords: esophagus cancer; radio-chemotherapy; ESD
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — pathological tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prophylactic chemoradiotherapy: pT1a -MM and pT1b-SM1 without pathological risk factors
  Interventions: Radiation: chemo-radiation
- Intensive chemoradiotherapy: pT1b-SM2; pT1a -MM and pT1b-SM1 with pathological risk factors
  Interventions: Radiation: chemo-radiation
- Radical chemoradiotherapy: Positive vertical margin or unknown margin
  Interventions: Radiation: chemo-radiation

INTERVENTIONS:
Radiation: chemo-radiation — different Chemo-radiotherapy regimen

SUMMARY:
This multicenter, prospective observational cohort study has the potential to optimize individualized chemoradiotherapy regimen for early-stage esophageal cancer patients who have received endoscopic submucosal dissection.

DETAILED DESCRIPTION:
Our study can further improve the local-regional lymph nodes control rate and alleviate the toxicity of chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Esophageal cancer patients who are pathologically confirmed as pT1a-MM stage or pT1b stage after endoscopic submucosal dissection； 2. No definite contraindications for chemo-radiotherapy； 3. Informed consent has been signed； 4. Refused surgery after endoscopic submucosal dissection.

Exclusion Criteria:

* 1. Severe heart, brain, lung disease or renal dysfunction; 2. Previous history of other malignancies; 3. Prior radiation or chemotherapy 4. Researchers consider it inappropriate to participate in this experiment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer patients, and pathologic-comfirmed pT1a-MM stage or pT1b stage
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxic events | 2026.2
  esophageal stenosis, radiation pneumonitis, etc

SECONDARY OUTCOMES:
3-year overall survival | 2029.1
  the time from randomization until death from any cause
3-year local-regional recurrence free survival | 2029.1
  the time from randomization until local-regional recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xu, MD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou

IPD SHARING:
Plan to Share IPD: No